CLINICAL TRIAL: NCT01647334
Title: Shrinking Target Adaptive Radiotherapy for Locally Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Regional Cancer Program, Canada (Other)
Responsible Party: Principal Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lung-START
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Shrinking Target Adaptive Radiotherapy (Experimental): Shrinking Target Adaptive Radiotherapy for Locally Advanced Non-Small Cell Lung Cancer
  Interventions: Radiation: Adaptive radiotherapy

INTERVENTIONS:
Radiation: Adaptive radiotherapy

SUMMARY:
This study aims to use a type of radiation (adaptive radiotherapy) to deliver curative-intent treatment to patients with non-small cell lung cancer, whose tumors would otherwise be too large for standard curative treatment. The study will use adaptive radiotherapy to achieve these goals. Adaptive radiotherapy is a process whereby treatment plans are modified during the course of treatment due to patient and tumor variations (ie. weight loss or tumor shrinkage). This may allow for dose escalation, while limiting the side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* ECOG performance status 0-2
* Histologically confirmed non-small cell lung carcinoma
* Locally advanced stage IIIA or IIIB lung carcinoma according to AJCC 7th edition
* Expected lung V20 of 35-60%, as determined at the time of 4D-CT simulation
* Assessment by medical oncologist and radiation oncologist, with adequate hepatic and renal function for administration of cisplatin-based doublet chemotherapy, at the discretion of the medical oncologist

Exclusion Criteria:

* Serious medical comorbidities or other contraindications to radiotherapy or chemotherapy
* Prior history of lung cancer within 5 years
* Prior thoracic radiation at any time
* Metastatic disease
* in some select cases, patients with a solitary metastasis (i.e. brain metastasis) may receive radical chemoradiotherapy after resection/ablation of their metastatic lesion, as standard practice. In such cases, the patient may be enrolled onto this study at the discretion of the local principle investigator once the metastasis has been treated.
* inability to attend full course of radiotherapy of follow-up visits
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Tumor reduction | 2.5 years (end of treatment)

SECONDARY OUTCOMES:
Rate of tumor shrinkage | 2.5 years (end of treatment)
Change in lung dose | 2.5 years (end of treatment)
Delivered doses | 2.5 years (end of treatment)
Radiation pneumonitis rates | 6 months, 12 months, 18 months, 24 months, 30 months (semi-annually)
Local control | 2.5 years (end of treatment)
Overall survival | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, PhD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute
Locations (1):
- London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario, Canada